CLINICAL TRIAL: NCT03287531
Title: Effect of Conventional Therapy and Low Level Laser Therapy on Pain and Function in Patients
Brief Title: Effect of Conventional Therapy and Low Level Laser Therapy on Pain and Function in Patients With Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emad Eldin Mohamed (Other)
Responsible Party: Sponsor-Investigator, Emad Eldin Mohamed, Effect of conventional therapy and low level laser therapy on pain and function in patients with temporomandibular joint dysfunction, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00500
Record Dates: First submitted 2017-09-16; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Low Level Laser Therapy; Temporomandibular Joint Dysfunction
Keywords: conventional therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional therapy (group I) (Experimental): 1. Exercise therapy.
     For muscles around TMJ :
     Masetter Lateral Pterygoid Medial Pterygoid Temporalis Digastric
  2. Pulsed ultrasound at 0.3 to 0.6 watts per sq cm over the lateral poles of the temporomandibular joint condyles with a small sound head for 2 to 3 minutes per side
  Interventions: Other: conventional therapy; Other: low level laser therapy
- low level laser therapy (groupII) (Experimental): LLLT with the appropriate parameters (904 nm, 8 j/cm2, 250mw) for duration of 20 min with repletion of three treatment sessions per week.
  Interventions: Other: low level laser therapy

INTERVENTIONS:
Other: conventional therapy — Exercise therapeutic Ultrasound
  Other Names: I
  Arms: conventional therapy (group I)
Other: low level laser therapy — LLLT with the appropriate parameters (904 nm, 8 j/cm2, 250mw) for duration of 20 min with repletion of three treatment sessions per week.
  Other Names: II

SUMMARY:
This study was to determine the effect of conventional therapy and low level laser therapy on pain and function in patients with temporomandibular joint dysfunction. sixty patients with myofascial pain syndrome of TMJ are randomly classified into two groups with thirty patients in each group; Group I received traditional exercise. Group II received low level laser therapy in addition to traditional exercise. All outcome measures including Pain and function, were evaluated before and after the treatment program.

DETAILED DESCRIPTION:
METHODOLOGY

Subjects: This prospective study was conducted on thirty patients of both genders with myofascial pain syndrome of TMJ in the department of physical therapy at October 6 university Hospital from December 2016 to October 2017. The Patients were selected to be enrolled into this study according to the following criteria:

ELIGIBILITY:
Inclusion Criteria:

* All patients are diagnosed as myofascial pain syndrome of TMJ.

Exclusion Criteria:

* Presence of systematic musculo-articular pathologies.
* Pregnant women.
* History of facial trauma.
* Facial palsy.
* Fractures of the facial bones.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Pain algometry | 4 weeks

SECONDARY OUTCOMES:
Jaw Functional questionnaire | 4 weeks